CLINICAL TRIAL: NCT01984268
Title: Adenocorticotrophic Hormone for Acute Treatment of Rheumatoid Arthritis Patients With Inadequate Response to Methotrexate
Brief Title: ACTHAR for Acute Treatment of Rheumatoid Arthritis Patients With Inadequate Response to Methotrexate
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D13146
Record Dates: First submitted 2013-11-08; First posted 2013-11-14 (Estimated); Results first posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2020-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; ACTHAR; Methotrexate; Inadequate response
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Four week ACTHAR treatment (Experimental): Rheumatoid arthritis subjects with inadequate response to methotrexate will be randomized to receive twice a week dosing of ACTHAR for a period of four weeks.
  Interventions: Drug: ACTHAR
- Twelve week ACTHAR treatment (Experimental): Rheumatoid arthritis subjects with inadequate response to methotrexate will be randomized to receive twice a week dosing of ACTHAR for a period of twelve weeks.
  Interventions: Drug: ACTHAR

INTERVENTIONS:
Drug: ACTHAR
  Other Names: Corticotropin

SUMMARY:
Adenocorticotrophic Hormone provides safe and effective treatment to induce disease remission in rheumatoid arthritis patients with active disease due to an inadequate response to methotrexate.

DETAILED DESCRIPTION:
The standard treatment for rheumatoid arthritis is using disease-modifying anti-rheumatic drugs such as methotrexate to control joint pain and swelling. Often times rheumatoid arthritis patients experience inadequate response to methotrexate with acute or persistent joint pain and swelling. In these patients, alternative or additional immunosuppressive therapy is needed to induce disease remission. In the present clinical trial, ACTHAR is being studied to induce disease remission on rheumatoid arthritis patients who have inadequate response to methotrexate therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age at the time of screening
* Subject is diagnosed with RA no less than 6 months prior to the screening
* Subject meets the 2010 ACR/EULAR Classification Criteria for RA (Arthritis Rheum 2010:62;2569-2581) with a score of ≥6
* Subject is seropositive for RF and/or anti-CCP antibodies as part of the diagnostic criteria for RA
* Subject has moderately to severely active RA during screening, as defined by a DAS28-ESR > 3.2
* Subject has moderately to severely active RA defined as the presence of at least 6/68 tender joints and at least 6/66 swollen joints
* Subject has had an inadequate response to the continuous use of methotrexate for at least 12 weeks prior to study entry with a nonchanging dose for at least 8 weeks prior to study entry

Exclusion Criteria:

* Treatment with any investigational agent within 4 weeks (or 5 half-lives of the investigational drug, whichever is longer) of screening
* Treatment with any biological agents within 4 weeks (or 5 half-lives of the agent, whichever is longer) of screening
* Immunization with a live/attenuated vaccine within 4 weeks prior to baseline
* Evidence of serious uncontrolled concomitant cardiovascular, nervous system, pulmonary (including obstructive pulmonary disease), renal, hepatic, endocrine (including Cushing's disease or uncontrolled diabetes mellitus) or gastrointestinal disease (including complicated diverticulitis, ulcerative colitis, or Crohn's disease.)
* Current liver disease as determined by principal investigator unless related to primary disease under investigation
* Known active current or history of recurrent bacterial, viral, fungal, mycobacterial or other infections (including but not limited to tuberculosis and atypical mycobacterial disease, Hepatitis B and C, and herpes zoster, but excluding fungal infections of nail beds)
* Any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening
* Active TB requiring treatment within the previous 3 years. Patients should be screened for latent TB and, if positive, treated following local practice guidelines prior to initiating treatment. Patients treated for tuberculosis with no recurrence in 3 years are permitted.
* Evidence of active malignant disease, malignancies diagnosed within the previous 10 years (including hematological malignancies and solid tumors, except basal and squamous cell carcinoma of the skin or carcinoma in situ of the cervix uteri that has been excised and cured), or breast cancer diagnosed within the previous 20 years unless related to primary disease under investigation
* Pregnant women or nursing (breast feeding) mothers
* Patients with reproductive potential not willing to use an effective method of contraception.
* History of alcohol, drug or chemical abuse within 1 year prior to screening.
* Neuropathies or other conditions that might interfere with pain evaluation unless related to primary disease under investigation.
* Body weight of > 150 kg
* Serum creatinine > 1.6 mg/dL (141 µmol/L) in female subjects and > 1.9 mg/dL (168 µmol/L) in male subjects. Subjects with serum creatinine values exceeding limits may be eligible for the study if their estimated glomerular filtration rates (GFR) are >30
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 1.5 times upper limit of normal (ULN)
* Total Bilirubin > ULN
* Platelet count < 100 x 109/L (100,000/mm3)
* Hemoglobin < 85 g/L (8.5 g/dL; 5.3 mmol/L)
* White Blood Cells < 3.0 x 109/L (3000/mm3)
* Absolute Neutrophil Count < 2.0 x 109/L (2000/mm3)
* Absolute Lymphocyte Count < 0.5 x 109/L (500/mm3)
* Positive Hepatitis BsAg or Hepatitis C antibody
* Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following randomization
* A diagnosis of any of the followings: scleroderma, osteoporosis, infection throughout the body, ocular herpes simplex, history of or a current stomach ulcer, uncontrolled hypertension (systolic blood pressure greater than 160), or allergy to pig-derived proteins
* Subject does not tolerate methotrexate and/or NSAID due to side effects or toxicities

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-06-23; Primary Completion 2016-09-01 (Actual); Study Completion 2016-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard C Chou, MD PhD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Entire Study: The study was placed on voluntary hold prior to completion by the PI. The voluntary hold stayed in place until the study's IRB approval expired. The study was subsequently closed by the IRB. The PI no longer has access to any data, and the PI has left the institution. No reportable study outcome data is available as determined by the IRB.
Period: Overall Study
Arm/Group | Entire Study
Started | 15
Completed | 0
Not Completed | 15
Not completed — Study Terminated | 15

BASELINE CHARACTERISTICS:
Population: The study was placed on voluntary hold prior to completion by the PI. The voluntary hold stayed in place until the study's IRB approval expired. The study was subsequently closed by the IRB. The PI no longer has access to any data, and the PI has left the institution. No reportable study outcome data is available as determined by the IRB.
Arm/Group | Entire Study
Number analyzed (Participants) | 15
Age, Customized [Count of Participants; unit: Participants]
  >18 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Disease Activity as Measured by ACR20 and ACR50.
Time Frame: 36 weeks
Population: as for baseline characteristics
Arm/Group | Entire Study
Number analyzed (Participants) | 0

2. Secondary Outcome: Adverse Events
Time Frame: 36 weeks
Population: as for baseline characteristics
Arm/Group | Entire Study
Number analyzed (Participants) | 0

3. Other Pre Specified Outcome: Change From Baseline in the Health Assessment Questionnaire Disability Index (HAQ-DI)
Time Frame: 36 weeks
Population: as for baseline characteristics
Arm/Group | Entire Study
Number analyzed (Participants) | 0

4. Other Pre Specified Outcome: Change From Baseline in the Short Form-36 (SF-36) Item Questionnaire Physical Component Summary (PCS)
Time Frame: 36 weeks
Population: as for baseline characteristics
Arm/Group | Entire Study
Number analyzed (Participants) | 0

5. Other Pre Specified Outcome: Change From Baseline in the Short Form-36 (SF-36) Item Questionnaire Mental Component Summary (MCS)
Time Frame: 36 weeks
Population: as for baseline characteristics
Arm/Group | Entire Study
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Change From Baseline in Patient's Assessment of Arthritis Pain - Visual Analog Scale (VAS)
Time Frame: 36 weeks
Population: as for baseline characteristics
Arm/Group | Entire Study
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The study was placed on voluntary hold prior to completion by the PI. The voluntary hold stayed in place until the study's IRB approval expired. The study was subsequently closed by the IRB. The PI no longer has access to any data, and the PI has left the institution. No reportable study outcome data is available as determined by the IRB.
Description: The study was placed on voluntary hold prior to completion by the PI. The voluntary hold stayed in place until the study's IRB approval expired. The study was subsequently closed by the IRB. The PI no longer has access to any data, and the PI has left the institution. No reportable study outcome data is available as determined by the IRB.
Arm/Group | Entire Study
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No